CLINICAL TRIAL: NCT04644120
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of ABBV-47D11 and ABBV-2B04 as Monotherapy or Combination Therapy in Adults With COVID-19
Brief Title: Study to Assess Adverse Events and How Intravenous (IV) ABBV-47D11 and IV ABBV-2B04 Given Alone and in Combination Moves Through the Body of Adult Participants With Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M20-404; 2020-005203-39 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-11-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: CoronaVirus Disease-2019 (COVID-19)
Keywords: CoronaVirus Disease-2019; COVID-19; Severe Acute Respiratory Syndrome Coronavirus-2; SARS-CoV-2; ABBV-47D11; ABBV-2B04
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- Part A: Group 1: ABBV-47D11 Dose A (Experimental): Participants will receive ABBV-47D11 Dose A on Day 1.
  Interventions: Drug: ABBV-47D11
- Part A: Group 1: Placebo for ABBV-47D11 (Placebo Comparator): Participants will receive placebo for ABBV-47D11 on Day 1.
  Interventions: Drug: Placebo for ABBV-47D11
- Part A: Group 2: ABBV-47D11 Dose B (Experimental): Participants will receive ABBV-47D11 Dose B on Day 1.
  Interventions: Drug: ABBV-47D11
- Part A: Group 2: Placebo for ABBV-47D11 (Placebo Comparator): Participants will receive placebo for ABBV-47D11 on Day 1.
  Interventions: Drug: Placebo for ABBV-47D11
- Part A: Group 3: ABBV-47D11 Dose C (Experimental): Participants will receive ABBV-47D11 Dose C on Day 1.
  Interventions: Drug: ABBV-47D11
- Part A: Group 3: Placebo for ABBV-47D11 (Placebo Comparator): Participants will receive placebo for ABBV-47D11 on Day 1.
  Interventions: Drug: Placebo for ABBV-47D11
- Part B: Group 1: ABBV-2B04 Dose A (Experimental): Participants will receive ABBV-2B04 Dose A on Day 1.
  Interventions: Drug: ABBV-2B04
- Part B: Group 1: ABBV-2B04 Dose A + ABBV-47D11 (Experimental): Participants will receive ABBV-2B04 Dose A in combination with ABBV-47D11 on Day 1.
  Interventions: Drug: ABBV-47D11; Drug: ABBV-2B04
- Part B: Group 1: Placebo (Placebo Comparator): Participants will receive Placebo for ABBV-2B04 followed by Placebo for ABBV-47D11 on Day 1.
  Interventions: Drug: Placebo for ABBV-47D11; Drug: Placebo for ABBV-2B04
- Part B: Group 2: ABBV-2B04 Dose B (Experimental): Participants will receive ABBV-2B04 Dose B on Day 1.
  Interventions: Drug: ABBV-2B04
- Part B: Group 2: ABBV-2B04 Dose B + ABBV-47D11 (Experimental): Participants will receive ABBV-2B04 Dose B in combination with ABBV-47D11 on Day 1.
  Interventions: Drug: ABBV-47D11; Drug: ABBV-2B04
- Part B: Group 2: Placebo (Placebo Comparator): Participants will receive Placebo for ABBV-2B04 followed by Placebo for ABBV-47D11 on Day 1.
  Interventions: Drug: Placebo for ABBV-47D11; Drug: Placebo for ABBV-2B04

INTERVENTIONS:
Drug: ABBV-47D11 — Intravenous (IV) infusion.
  Arms: Part A: Group 1: ABBV-47D11 Dose A; Part A: Group 2: ABBV-47D11 Dose B; Part A: Group 3: ABBV-47D11 Dose C; Part B: Group 1: ABBV-2B04 Dose A + ABBV-47D11; Part B: Group 2: ABBV-2B04 Dose B + ABBV-47D11
Drug: Placebo for ABBV-47D11 — Intravenous (IV) infusion.
  Arms: Part A: Group 1: Placebo for ABBV-47D11; Part A: Group 2: Placebo for ABBV-47D11; Part A: Group 3: Placebo for ABBV-47D11; Part B: Group 1: Placebo; Part B: Group 2: Placebo
Drug: ABBV-2B04 — Intervenous (IV) Infusion
  Arms: Part B: Group 1: ABBV-2B04 Dose A; Part B: Group 1: ABBV-2B04 Dose A + ABBV-47D11; Part B: Group 2: ABBV-2B04 Dose B; Part B: Group 2: ABBV-2B04 Dose B + ABBV-47D11
Drug: Placebo for ABBV-2B04 — Intervenous (IV) Infusion
  Arms: Part B: Group 1: Placebo; Part B: Group 2: Placebo

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Lung failure is the main cause of death related to COVID-19 infection. The main objective of this study is to evaluate the safety and tolerability of ABBV-47D11 and ABBV-2B04 given alone and in combination to participants with COVID-19 infection. In addition, this study will evaluate the pharmacokinetics (how the body handles the study drug) and anti-viral activity of the study drug.

ABBV-47D11 and ABBV-2B04 are investigational anti-SARS-CoV-2 monoclonal antibodies being developed for the treatment of COVID-19. Study will be conducted in two parts. In part A, participants will receive ABBV-47D11 or placebo. There is a 1 in 4 chance that participants will be assigned to placebo. In part B, participants will receive ABBV-2B04 alone or in combination with ABBV-47D11 or placebo. There is a 1 in 5 chance that participants will be assigned to placebo. Around 54 adult participants with COVID-19 will be enrolled in approximately 10 to 30 sites globally.

In part A participants will receive single intravenous (into the veins) infusion of ABBV-47D11 or placebo on Day 1. In part B participants will receive single intravenous (into the veins) infusion of ABBV-2B04 alone or in combination with ABBV-47D11 or placebo on Day 1. Participants will be followed up for 106 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. The effect of the treatment will be checked by medical assessments, blood tests, nasal swabs and presence of side effects.

DETAILED DESCRIPTION:
Part B of this study was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 infection based on initial nucleic acid or antigen testing from respiratory swab, saliva, or other bodily fluid within 7 days prior to randomization.
* Must have >= 1 symptom associated with COVID-19 with an onset of <= 8 days prior to randomization.
* Hospitalized or plans for hospital admission due to COVID-19 at the time of randomization or not currently hospitalized and does not have plans for hospital admission at the time of randomization, but is willing to be confined for ≥ 48 hours post-dose for the purposes of participating in this research study

Exclusion Criteria:

* Have an oxygen saturation (SpO2) < 88% on room air at rest for 5 minutes OR ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <= 200 mmHg at randomization.
* Requiring high-flow nasal cannula oxygen therapy/non-invasive or invasive mechanical ventilation/extracorporeal membrane oxygenation (ECMO) or anticipated impending need for high-flow nasal cannula oxygen therapy/non-invasive or invasive mechanical ventilation/ECMO.
* Prior treatment with a SARS-CoV-2 specific monoclonal antibody or convalescent COVID-19 plasma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Study-Drug Related Grade 3 or Higher Adverse Events (AEs) | Up to Day 106
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug.
Number of Participants With Study-Drug Related Grade 3 or Higher Infusion-Related Reactions | Up to Day 106
  Participants will be assessed for the infusion-related reaction considered drug-related by the investigator.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of ABBV-47D11 | Up to Day 85
  Maximum observed serum concentration (Cmax) of ABBV-47D11.
Time to Cmax (Tmax) of ABBV-47D11 | Up to Day 85
  Time to maximum serum concentration of ABBV-47D11.
Area Under the Serum Concentration-Time Curve (AUC) From Day 1 (0 hour) to Day 29 (672 hour) (AUC0-672h) of ABBV-47D11 | Up to Day 29
  Area Under the Serum Concentration-Time Curve (AUC) From Day 1 (0 hour) to Day 29 (672 hour) (AUC0-672h) of ABBV-47D11.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-47D11 | Up to Day 85
  Terminal phase elimination half-life (t1/2) of ABBV-47D11.
AUC From Time 0 to Infinity (AUCinf) of ABBV-47D11 | Up to Day 85
  AUC From Time 0 to Infinity (AUCinf) of ABBV-47D11.
Detection of Anti-Drug Antibodies (ADA) for ABBV-47D11 | Up to Day 85
  Anti-drug antibodies will be detected using a tiered approach for ABBV-47D11.
Detection of Neutralizing Anti-Drug Antibodies (nADA) for ABBV-47D11 | Up to Day 85
  Neutralizing anti-drug antibodies will be detected using a tiered approach for ABBV-47D11.
AUC for Change From Baseline (Day 1) in SARS-CoV-2 Ribose Nucleic Acid (RNA) Reverse Transcription-Polymerase Chain Reaction (RT-PCR) | Baseline (Day 1) through Day 29
  Area Under the Serum Concentration-Time Curve (AUC) of SARS-CoV-2 RNA.
Time to Negative SARS-CoV-2 by RT-PCR | Up to Day 29
  Number of days from Baseline (Day 1) to negative SARS-CoV-2 by RT-PCR.
Negative SARS-CoV-2 RNA by RT-PCR | Up to Day 15
  Number of participants with negative SARS-CoV-2 RNA by RT-PCR.
Maximum Observed Serum Concentration (Cmax) of ABBV-2B04 | Up to Day 85
  Maximum observed serum concentration (Cmax) of ABBV-2B04.
Time to Cmax (Tmax) of ABBV-2B04 | Up to Day 85
  Time to maximum serum concentration of ABBV-2B04.
Area Under the Serum Concentration-Time Curve (AUC) From Day 1 (0 hour) to Day 29 (672 hour) (AUC0-672h) of ABBV-2B04 | Up to Day 29
  Area Under the Serum Concentration-Time Curve (AUC) From Day 1 (0 hour) to Day 29 (672 hour) (AUC0-672h) of ABBV-2B04.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-2B04 | Up to Day 85
  Terminal phase elimination half-life (t1/2) of ABBV-2B04.
AUC From Time 0 to Infinity (AUCinf) of ABBV-2B04 | Up to Day 85
  AUC From Time 0 to Infinity (AUCinf) of ABBV-2B04.
Detection of Anti-Drug Antibodies (ADA) for ABBV-2B04 | Up to Day 85
  Anti-drug antibodies will be detected using a tiered approach for ABBV-2B04.
Detection of Neutralizing Anti-Drug Antibodies (nADA) for ABBV-2B04 | Up to Day 85
  Neutralizing anti-drug antibodies will be detected using a tiered approach for ABBV-2B04.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- United States (11):
  - Glendale Adventist Medical Center /ID# 225188, Glendale, California
  - Beautiful Minds Clinical Research Center /ID# 228708, Cutler Bay, Florida
  - University of Miami /ID# 225038, Miami, Florida
  - Triple O Research Institute /ID# 228612, West Palm Beach, Florida
  - University of Illinois Hospital and Health Sciences System /ID# 224323, Chicago, Illinois
  - Pikeville Medical Center /ID# 224539, Pikeville, Kentucky
  - Saint Peter's University Hospital /ID# 225183, New Brunswick, New Jersey
  - Saint Michael's Medical Center /ID# 225258, Newark, New Jersey
  - The Christ Hospital /ID# 224541, Cincinnati, Ohio
  - Prisma Health Children's Hospital Upstate /ID# 224556, Greenville, South Carolina
  - Gadolin Research, LLC /ID# 229394, Beaumont, Texas
- Hungary (2):
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz /ID# 226015, Budapest
  - Semmelweis Egyetem /ID# 226016, Budapest
- Israel (2):
  - Hadassah Medical Center-Hebrew University /ID# 225827, Jerusalem
  - Sheba Medical Center /ID# 225857, Tel Hashomer, Ramat Gan
- Universitair Medisch Centrum Utrecht /ID# 225919, Utrecht, Netherlands
- Puerto Rico (2):
  - San Juan Bautista School of Medicine /ID# 225963, Caguas
  - Manati Medical Center /ID# 225936, Manatí

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343